CLINICAL TRIAL: NCT02700893
Title: Cerebral NIRS Profiles During Premedication for Neonatal Intubation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other); Centre de Recherche Clinique du CHIC (Unknown)
Responsible Party: Principal Investigator, Xavier Durrmeyer, MD, PhD, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRETTINEO sub-study
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Premedication; Endotracheal Intubation; Cerebral Hypoperfusion
MeSH Terms: interventions — Atropine; Atracurium; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atropine + propofol (Experimental): Atropine bolus: 20 µg/kg Propofol injected over 60 seconds: 1 mg/kg for infants < 1000g - Renewable once 2.5 mg/kg for infants > 1000G - Possible additional dose of 1 mg/kg
  Interventions: Drug: atropine+ propofol
- Atropine + atracurium + sufentanil (Active Comparator): Atropine bolus: 20 µg/kg Atracurium: 0.3 mg/kg- Possible additional dose of 0.1 mg/kg Sufentanil: 0.1 µg/kg for infants < 1000g 0.2 µg/kg for infants > 1000g
  Interventions: Drug: atropine + atracurium + sufentanil

INTERVENTIONS:
Drug: atropine+ propofol — Atropine bolus: 20 µg/kg Propofol injected over 60 seconds: 1 mg/kg for infants < 1000g - Renewable once 2.5 mg/kg for infants > 1000G - Possible additional dose of 1 mg/kg
  Arms: Atropine + propofol
Drug: atropine + atracurium + sufentanil — Atropine bolus: 20 µg/kg Atracurium: 0.3 mg/kg- Possible additional dose of 0.1 mg/kg Sufentanil: 0.1 µg/kg for infants < 1000g 0.2 µg/kg for infants > 1000g
  Arms: Atropine + atracurium + sufentanil

SUMMARY:
Observational ancillary study of the PRETTINEO study (ClinicalTrials.gov Identifier: NCT01490580) which is a multicenter double blind randomized controlled trial comparing "atropine+propofol" vs "atropine+atracurium+sufentanil" as a premedication prior to endotracheal intubation of the neonate.

Primary outcome:

* Cerebral desaturation defined by a rScO2 delta >20% from the baseline value (before premedication).
* Variation of more than 10% of cerebral FTOE (Fractional Tissue Oxygen Extraction) during premedication, calculated from rScO2 and pulse oximetry with the formula FTOE=SaO2 - rScO2/SaO2 .

Hypothesis: "atropine + propofol" compared to "atropine+atracurium+sufentanil" does not increase the frequency of cerebral hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Corrected age < 45 weeks of gestational age
* Currently hospitalized in a neonatal intensive care unit
* Requiring semi-urgent or elective intubation
* Equipped with a reliable and permeable IV line
* Parental consent

Exclusion Criteria:

* Lack of parental consent
* Parental refusal
* Sedative or anesthetic treatment in the previous 24 hours
* Hemodynamic compromise defined as mean blood pressure< corrected GA and/or refill time > 3 seconds
* Upper airway malformation
* Life-threatening situation requiring immediate intubation
* Inclusion in another trial not permitting any other participation
* Impossibility to establish venous access
* Any contra-indication to any experimental drug
* Skin lesions or burns of the forehead

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cerebral desaturation | from 1 minute before to 60 minutes after the start of premedication
  rScO2 delta >20% from the baseline value (before premedication). rScO2 recording measured by INVOS 1500C 1 minute before the first injection and at 3, 6, 9, 12, 15, 30, 45 and 60 minutes after the first drug injection
FTOE (Fractional Tissue Oxygen Extraction) | from 1 minute before to 60 minutes after the start of premedication
  Variation of more than 10% of cerebral FTOE (Fractional Tissue Oxygen Extraction) during premedication. FTOE is calculated from rScO2 and pulse oxymetry (SaO2) with the formula FTOE = SaO2 - rScO2/SaO2. Values will be recorded
  1 minute before the first injection and at 3, 6, 9, 12, 15, 30, 45 and 60 minutes after the first drug injection.

CONTACTS AND LOCATIONS:
Overall Officials: Meryl Vedrenne-Cloquet, MD, Principal Investigator — CHI Créteil; Xavier Durrmeyer, MD, PhD, Study Director — CHI Créteil
Locations (2):
- France (2):
  - Hôpital intercommunal de Créteil, Créteil
  - Hôpital des enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vedrenne-Cloquet M, Breinig S, Dechartres A, Jung C, Renolleau S, Marchand-Martin L, Durrmeyer X. Cerebral Oxygenation During Neonatal Intubation-Ancillary Study of the Prettineo-Study. Front Pediatr. 2019 Mar 1;7:40. doi: 10.3389/fped.2019.00040. eCollection 2019. PMID 30881948
- See also: Open access article — https://www.frontiersin.org/articles/10.3389/fped.2019.00040/full